CLINICAL TRIAL: NCT01575470
Title: Treatment of Severe Adult Traumatic Brain Injury Using Bone Marrow Mononuclear Cells
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Charles Cox, Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-11-0477; Award No. W81XWH-11-1-0460 (Other: USAMRMC)
Record Dates: First submitted 2012-04-06; First posted 2012-04-11 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury; TBI; stem cells
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- bone marrow mononuclear cells (Experimental): a bone marrow harvest will be performed within 36 hours of injury followed by a single intravenous infusion of autologous bone marrow mononuclear cells (BMMNCs)
  Interventions: Biological: autologous bone marrow mononuclear cells

INTERVENTIONS:
Biological: autologous bone marrow mononuclear cells — bone marrow harvest (5ml/kg of body weight) performed within 36 hours of injury, followed by single intravenous infusion of bone marrow mononuclear cells.
  Other Names: BMMNCs

SUMMARY:
The purpose of this study is to determine if bone marrow harvest, BMMNC separation, and re-infusion in adults with acute severe TBI is safe and will improve functional outcome.

12/09/2015 Update: The study is closed to new enrollment and all follow-up visits have been completed. Data analysis is underway.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) contributes to 50% of all trauma deaths. The mortality rate for adults following severe TBI (Glasgow Coma Scale < 9) is estimated to be 33%. There is currently no therapy to reverse the primary injury associated with TBI. Over the past 10 years there has been a growing body of literature supporting the use of various progenitor cell types to treat acute neurological injuries such as TBI and stroke. Neural stem cells (adult and embryonic), mesenchymal stromal and multipotent adult progenitor cells, and bone marrow mononuclear cells (from which MSC and MAPCs are derived) have all shown efficacy in pre-clinical models of TBI/stroke through various mechanisms; however, few groups believe that true neural replacement and integration are the putative mechanisms involved in the observed efficacy. More likely is that the progenitor cell populations are modifying the regional response to injury (inflammatory/reparative vs. regenerative), resulting in improved functional outcomes. Our primary hypothesis is that bone marrow mononuclear cell (BMMNC) autologous transplantation after TBI is safe (harvest and infusion related toxicity) after TBI. Our secondary hypothesis is that functional outcomes measures will improve after BMMNC infusion, (3) BMMNC infusion will reduce BBB permeability, (4) BMMNC is neuroprotective and preserves grey matter and white matter volumes after TBI.

Patients, ages18 to 55 years old, admitted to Memorial Hermann Hospital Trauma Center with Glasgow Coma Scores (GCS) of 5 to 8 will be screened. Those patients meeting inclusion/exclusion criteria (or their Legal Authorized Representative [LAR]) will be offered consent to participate. This is a dose-escalation study consisting of 4 cohorts including a control group (5 subjects/cohort). The first five subjects will not undergo the bone marrow harvest procedure; though they will be followed and treated the same as the other study participants and complete all follow-up procedures. Subjects 6-10 will receive the lowest dose target of 6X106 mononuclear cells/kilogram body weight. Subjects 11-15 will receive 9x106 mononuclear cells/kilogram body weight, and lastly Subjects 16-20 will receive 12X106 mononuclear cells/kilogram body weight. The study is NOT powered to detect functional measures of efficacy. However, estimates can be made regarding potential treatment effect sizes to allow rational power analyses for the follow-on Phase II study. This study should determine if bone marrow harvest, BMMNC separation, and reinfusion is safe in adults with acute, severe TBI.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 55 years of age on the day of injury;
* Hospital admission Glasgow Coma Score between 5 and 8;
* Initial injury occurring less than 24 hours prior to consent;
* Ability to speak English.

Exclusion Criteria:

* Known history of:

  1. brain injury,
  2. psychiatric disorder,
  3. neurological impairment and/or deficit
  4. seizure disorder requiring anti-convulsant therapy
  5. recently treated infection
  6. renal disease or altered renal function
  7. hepatic disease or altered liver function
  8. cancer
  9. substance abuse of positive urine drug screen at admission
  10. immunosuppression
  11. HIV
* Obliteration of perimesencephalic cistern on initial head CT suggesting prolonged hypoxic ischemic insult
* Initial hospital ICP > 40mm Hg
* Hemodynamic instability at the time of consent defined as ongoing fluid resuscitation and/or requirement for inotropic support to maintain MAP at or above normals for age - does not include CPP based inotropic support
* Uncorrected coagulopathy at the time of bone marrow harvest defined as INR >1.6, PTT >36 sec, PLT < 100,000, Fibrinogen < 100g/dL
* Unstable pelvic fractures defined as requiring operative fixation to manage
* Pulmonary contusions defined as a chest x-ray with non-anatomic opacification and/or PaO2:FIO2 ratio < 250 associated with the mechanism or injury
* Greater than AAST Grade I solid or hollow visceral injury of the abdomen and/or pelvis as diagnosed by CT or other imaging
* Spinal cord injury as diagnosed by CT or MR imaging or clinical findings
* Persistent hypoxia defined as SaO2 < 94% for > 30 minutes occurring at any time from hospital admission to time of consent
* Weight > 300 lbs
* Any contraindication to MRI (including being too large to fit into the MRI)
* Positive urine pregnancy test
* Participation in a concurrent intervention study
* Unwillingness to return for follow-up visits

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2012-03; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
neurological events (seizures, changes in Glasgow coma score [GCS], cerebral vascular accident [CVA}) | 12 hours post product infusion up to 21 days post infusion

SECONDARY OUTCOMES:
infectious morbidity | up to 21 days post infusion
global functional status per the GOS-E | up to 6 months post injury/treatment
  the Glasgow Outcome Scale-Extended (GOS-E) will be administered to assess global functional status (consciousness, independence, work status, return of lifestyle)
global functioning per the Disability Rating Scale | up to 6 months post injury/treatment
  the Disability Rating Scale (DRS) will be administered which measures level of arousal, cognitive ability related to activities of daily living, motor response, feeding, toileting, grooming and employability

CONTACTS AND LOCATIONS:
Overall Officials: Charles S Cox, Jr., M.D., Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States